CLINICAL TRIAL: NCT00920010
Title: Lung Cancer Specimen Repository Protocol, Ancillary
Brief Title: S9925: Collecting and Storing Samples From Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000078624; S9925 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fixed tissue in paraffin blocks or slides, slides of buccal brushings, fresh frozen tissue peripheral blood, serum, plasma, white blood cells, and sputum.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: biologic sample preservation procedure

SUMMARY:
RATIONALE: Collecting and storing samples of tissue, blood, and sputum from patients with cancer to study in the laboratory may help the study of cancer in the future.

PURPOSE: The purpose of this study is to collect and store tissue, blood, and sputum samples from patients with lung cancer to be tested in the laboratory.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish a central lung cancer specimen repository to serve as a resource for current and future scientific studies.
* Correlate clinicopathologic information in the Southwest Oncology Group clinical data base with results of studies using the repository.
* Test new hypotheses with the specimens in the repository.

OUTLINE: Peripheral blood, sputum, and biopsy specimens are collected from patients. Tissue samples are frozen and stored in a lung cancer specimen repository for later use in correlative studies.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled on one of the following Southwest Oncology Group protocols:

  * SWOG-8805, SWOG-9019, SWOG-9416, SWOG-9509, SWOG-S9900, SWOG-S0003, SWOG-S0023, SWOG-S0126, SWOG-S0435, SWOG-S0220, SWOG-S0222, SWOG-S0327, SWOG-S0310, SWOG-S0339, SWOG-S0342, SWOG-S0341, SWOG-S0509, SWOG-S0429, or SWOG-S0124

PATIENT CHARACTERISTICS: Not specified

PRIOR CONCURRENT THERAPY: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung cancer patients registered to SWOG lung protocols.
Sampling Method: Non-Probability Sample
Enrollment: 2264 (Actual)
Dates: Start 2000-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Establishment of a central lung cancer specimen repository to serve as a resource for current and future scientific studies | From date of study activation to consolidation of specimen banks
Correlation of clinicopathologic information in the Southwest Oncology Group clinical data base with results of studies using the repository | From date of study activation to consolidation of specimen banks
Test of new hypotheses with the specimens in the repository | From date of study activation to consolidation of specimen banks

CONTACTS AND LOCATIONS:
Overall Officials: Wilbur A. Franklin, MD, Study Chair — University of Colorado, Denver
Locations (431):
- United States (431):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Highlands Oncology Group - Springdale, Bentonville, Arkansas
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Washington Township Hospital, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Mid-Illinois Hematology-Oncology Associates at Community Cancer Center, Normal, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - MaineGeneral Medical Center - Waterville, Waterville, Maine
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Winthrop University Hospital, Mineola, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming